CLINICAL TRIAL: NCT00509600
Title: Phase IIA Window Study of Etanercept (Enbrel) for Juvenile Myelomonocytic Leukemia
Brief Title: Etanercept (Enbrel) for Juvenile Myelomonocytic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment; study terminated.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0215
Record Dates: First submitted 2007-07-27; First posted 2007-07-31 (Estimated); Results first posted 2010-12-02 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Leukemia
Keywords: Juvenile Myelomonocytic Leukemia; JMML; Leukemia; Etanercept; Enbrel
MeSH Terms: conditions — Leukemia; Leukemia, Myelomonocytic, Juvenile | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Etanercept (Experimental): 0.8 mg/kg subcutaneously weekly for 90 days
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — 0.8 mg/kg Subcutaneously Once A Week for 90 Days
  Other Names: Enbrel

SUMMARY:
Primary Objectives:

1.1 Estimate rate of response and define acute toxicity to etanercept used in an up-front phase II window in newly diagnosed or relapsed JMML.

1.2 Determine if response to Tumor Necrosis Factor (TNF) blockade correlates with genetic basis of Juvenile Myelomonocytic Leukemia (JMML) [mutations in NF1, Ras, SHP2] or levels of TNFa.

1.3 Determine if TNF blockade by etanercept results in inhibition of free levels of TNFa and other cytokines by ELISA and bioassay and improves blood counts.

1.4 Estimate the two year event free survival and overall survival in JMML patients following etanercept and allogeneic hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
Etanercept blocks a hormone called Tumor Necrosis Factor (TNF), which has been shown to play a role in helping the growth of leukemic cells in JMML.

Before participants can start treatment on this study, they will have what are called "screening tests". These tests will help the doctor decide if patients are eligible to take part in the study. You will have a complete medical history and physical exam. About two tablespoons of blood and urine will be collected for routine tests as well as to test for the liver and kidney function. You will have a bone marrow biopsy performed to monitor disease activity. To collect a bone marrow biopsy, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow and bone is withdrawn through a large needle. You will have cells from inside of the mouth tested for genetic changes by swabbing the side of the cheeks.

If you are found to be eligible, etanercept will be given as an injection under the skin once a week for up to 90 days.

During the study, you will have weekly follow-up tests that will include physical exam and lab tests. About 2 tablespoons of blood will be collected each time. Urine will also be collected for testing at least every 3 weeks while on the study.

If the disease gets worse or intolerable side effects occur, you will be taken off study and alternative treatment options will be discussed.

This is an investigational study. The FDA has approved etanercept for use in adults and children with rheumatoid arthritis and juvenile rheumatoid arthritis. Its use in this study is experimental. A total of up to 30 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All children greater than 6 months of age and less than 18 years of age with newly-diagnosed previously untreated or previously diagnosed JMML, which has reoccurred after treatment with chemotherapy, stem cell transplantation, and/or cis-retinoic acid.
2. A diagnosis of JMML is confirmed only if the following criteria for JMML are met: a) ALL of the following: Absence of t(9;22) or BCR-ABL by PCR or FISH; Absolute monocyte count >1000 (1 X 109/µL); <20% bone marrow blasts; b) At least 2 of the following: Elevated Hb F hemoglobin; Myeloid precursors in peripheral blood; WBC >10,000 (10 X 109/µL); GM-CSF hypersensitivity in methylcellulose culture of bone marrow progenitors cells.
3. Adequate hepatic function (bilirubin equal or less than 2.0 mg/dl; ALT equal or less than 3x normal)
4. Adequate renal function (serum creatinine equal or less than 2 x normal)
5. Performance Status: Have a Karnofsky score >50.
6. Written, informed consent according to institution guidelines.

Exclusion Criteria:

1. Pregnant or lactating.
2. Receiving any other chemotherapy. Patients must have been off chemotherapy for at least 2 weeks and must have recovered from acute toxicity of all previous therapy prior to enrollment.
3. Febrile neutropenia at study entry.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2004-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Wells, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD . Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 05/19/04 through 03/05/09. All participants recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Study was terminated due to low accrual.
Period: Overall Study
Arm/Group | Etanercept
Started | 1
Completed | 0
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Etanercept
Number analyzed (Participants) | 1
Age Continuous [Mean (Full Range); unit: years] | 3 [3 to 3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Patient Response
Description: Response is defined as a WBC < 15,000 and platelets > 75,000 at 12 weeks; toxicity is defined as a grade 3 or worse infection or non-hematologic toxicity within the first 4 weeks.
Time Frame: 12 weeks
Population: No analysis as only registrant inevaluable, and trial terminated early due to poor enrollment.
Arm/Group | Etanercept
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Study period 4 years and 10 months. Only patient registered on study for two (2) months.
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept (N=1)
Toxicity (General disorders) | 1 (1) — Grade 3 Non-hematological Toxicity.

LIMITATIONS AND CAVEATS:
Early termination due to low accrual. Rare disease with less than 100 cases diagnosed per year.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No